CLINICAL TRIAL: NCT06660615
Title: The Effect of Midwife-Led Care on Perception of Labour Pain, Duration of Labour, Comfort of Labour and Respectful Maternity Care: A Single Blinded Randomised Controlled Trial
Brief Title: The Effect of Continuous Midwifery-led Care in Birth Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/1191
Record Dates: First submitted 2024-10-17; First posted 2024-10-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain
Keywords: Labour Pain; Respectful Motherhood Care; Birth Duration; Comfort of Birth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which group they are in, so they will be blind to differences in the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receiving midwife-led care (Experimental): The birth process will be followed by the same midwife from the beginning of the intrapartum period until the birth of the baby and placenta. In this process, positive respectful maternal care will be included in line with the recommendations of WHO (İsbir & Sercekuş, 2017).
  Interventions: Behavioral: MIDWIFE-LED CARE
- Midwife-Led Non-Care Receiving Care (No Intervention): Participants in the group will receive routine care normally provided only in the hospital. Within this care, from the beginning of the intrapartum period until the birth of the baby and placenta, the birth process will be followed under the supervision of a midwife or physician who is randomly available within the working conditions of the birth unit.

INTERVENTIONS:
Behavioral: MIDWIFE-LED CARE — The birth process will be followed by the same midwife from the beginning of the intrapartum period until the birth of the baby and placenta. In this process, positive respectful maternal care will be included in line with the recommendations of WHO (İsbir & Sercekuş, 2017).
  Arms: Receiving midwife-led care

SUMMARY:
Caesarean section is an emergency procedure necessary to prevent harm or death to the mother or newborn. Worldwide, caesarean section rates are steadily increasing. This increase not only has negative consequences on maternal and child health, but also leads to a reduction in essential resources and impedes access to health services worldwide. The International Federation of Gynaecology and Obstetrics (FIGO) has called for help from government bodies, professional organisations, women's groups and other stakeholders to reduce unnecessary caesarean sections. According to a review of antenatal and intrapartum interventions to reduce caesarean section, promote vaginal birth and reduce fear of childbirth; the importance of support in the intrapartum period is prominent. The National Institute for Health and Care Excellence (NICE) states that this support with a midwife who provides care and one-to-one support to the woman in labour reduces women's anxiety and increases their sense of trust.

DETAILED DESCRIPTION:
Vaginal delivery of low-risk pregnancies is best provided and guided by a midwife. It is seen that receiving support from a midwife in the birth of low-risk pregnancies does not increase the risks for the mother or newborn and has many economic and emotional advantages. The World Health Organisation recommends respectful care based on woman-centred care in the intapartum period for a positive birth experience. Respectful Maternity Care has been recognised as a key strategy to improve the quality of maternity care. Although there is no clear consensus on the definition of respectful maternity care, it is generally considered synonymous with intimate and woman-centred care. It is a care approach that emphasises the fundamental rights of women, newborns and families and increases adequate access to evidence-based care while recognising their needs and preferences. In this direction, midwives are expected to add respectful maternity care to their clinical skills in the management of the birth process. In the literature, it is seen that respectful and helpful interaction between women and health professionals during labour creates positive perceptions in women. In the study of Liu et al. (2021), it is stated that midwife-led management of labour leads to the formation of positive perceptions in women. Fear of labour, labour pain and duration of labour in midwife-led care on the behaviour of the students in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with spontaneous pregnancy between 38-42 weeks of gestation
* single fetus head presentation
* first pregnancy
* without any pregnancy-related risk status (such as preeclampsia, gestational diabetes)
* who were admitted to the delivery room for normal labour will be included in the study.

Exclusion Criteria:

* WOMEN WHO CANNOT GIVE BIRTH NORMALLY
* WANT TO LEAVE THE LABOUR FORCE

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — WOMEN IN LABOUR
Enrollment: 85 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
The Effect of Midwife-Led Care on Perception of Labour Pain, Duration of Labour, Comfort of Birth and Respectful Maternity Care | 1 years
  Measurement Tools Information Form (IF) (Appendix 1): This form was prepared in line with the literature (Liu et al., 2021) and includes socio-demographic and obstetric characteristics of the participants.
Birth Pain | 1 years
  Visual Analog Scale (VAS) (ANNEX-2): The Visual Analog Scale (VAS) was developed by Price et al. in 1983 and is used to measure pain intensity and for pain monitoring. The VAS is 10 cm long and the two ends are named differently. On the scale, '0' indicates no pain and '10' indicates the most severe level of pain. The VAS is a measurement tool that is frequently and reliably used to assess labor pain (Price et al., 1983; Mutlu & Özkaya, 2021).
birth monitoring | 1 years
  Birth Monitoring Form (DIF) (ANNEX-3) : It was aimed to evaluate the labour process with the labour monitoring form developed by the researchers. In the birth follow-up form, data obtained from pregnant women in G1 and G2 regarding cervical dilatation and dilatation, duration, frequency and intensity of contractions, time of delivery, and time of placental separation will be recorded.
Comfort of Birth | 1 years
  Birth Comfort Scale (BCS) (ANNEX-4): It was developed by Kerri Durnell Schuiling in 2003, inspired by Kolcaba's comfort theory. The original version consists of fourteen items. The scale is a five-point Likert-type scale (1= Strongly disagree, 5= Strongly agree). Its Turkish validity and reliability was performed by Potur et al. There are three subscales/factors (environmental, physical, psychospiritual) in the Turkish version of the comfort of labour scale consisting of nine items. Items 2,3,4,6 of the scale are divided into sub-dimensions in the physical dimension, items 7,8 in the psychospiritual dimension and items 1,5,9 in the environmental dimension. A minimum of 9 and a maximum of 45 points can be obtained from the scale. The Cronbach Alpha value of the scale was found to be 0.75 (Potur et al., 2015).

SECONDARY OUTCOMES:
Respectful Maternity Care | 1 years
  Respectful Motherhood Care Scale (RMCS) (ANNEX-5): The scale was developed by Dişsiz et al. in 2023. With the five-point Likert-type scale, it was aimed to evaluate the respectful maternity care perceived by women between the 6th week and 1 year postpartum during pregnancy, birth and postpartum period. The scale consists of a total of 29 items and 3 sub-dimensions with mixed positive and negative statements. The sub-dimensions are 'Consensual Dignified Care (17 items)', 'Psychological Abuse and Care Neglect (7 items)' and 'Physical Violence, Privacy Violation and Discrimination (5 items)'. The highest total score that can be obtained from the scale is 145 and the lowest score is 29. An increase in the score obtained from the overall scale indicates that the woman's perception that she received respectful maternity care during pregnancy, birth and postpartum period increased, while a decrease indicates that the woman's perception that she received respectful maternity care during pregn

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Nusaybi̇N State Hospital, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'm not sure right now.

REFERENCES:
- [Background] Visser GHA, Ayres-de-Campos D, Barnea ER, de Bernis L, Di Renzo GC, Vidarte MFE, Lloyd I, Nassar AH, Nicholson W, Shah PK, Stones W, Sun L, Theron GB, Walani S. FIGO position paper: how to stop the caesarean section epidemic. Lancet. 2018 Oct 13;392(10155):1286-1287. doi: 10.1016/S0140-6736(18)32113-5. No abstract available. PMID 30322563